CLINICAL TRIAL: NCT05300880
Title: Nursing Capacity Building in Health Coaching With Hospitalised Chronic Heart Failure Patients: An Intervention Study
Brief Title: Health Coaching With Hospitalised Chronic Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: HCHCHF
Record Dates: First submitted 2022-03-04; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-02

CONDITIONS: Education, Nursing
Keywords: Health coaching; Intervention; Chronic heart failure; Empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Training program — A multi-component intervention based on health coaching. The strategies of this program consisted in five 16-hour sessions using case studies to find out whether nurses were able to empower chronic cardiac patients and debriefing and a 4-hour booster session seven months later.

SUMMARY:
Background: Nurses, the usual leaders in the follow-up of chronic cardiac patients, need to improve their training so that they are in the best position to empower these patients. From this approach, health coaching is presented as an innovative and valid alternative. Despite this, no studies have been found that implement and evaluate this type of program in the hospital setting.

Purpose: to evaluate the preliminary efficacy of this programme for the development of nursing capacity in health coaching with CHF (Chronic Heart Failure) inpatients.

Method: An exploratory pre-post quasi-experimental pilot study. Nineteen nurses, the total population of nurses working in the cardiology ward, were recruited in September 2020. All the nurses received a multi-component intervention based on health coaching. The strategies of this program consisted in five 16-hour sessions using case studies to find out whether nurses were able to empower chronic cardiac patients and debriefing and a 4-hour booster session seven months later. The I-CEpSE instrument was used to assess outcomes. The primary outcome was the difference in the median of knowledge, skills and attitudes pre and post intervention (between T0-T1, T2-T3 and T0-T3). Changes within nurses were analyzed using U Mann-Whitney test for independent samples.

DETAILED DESCRIPTION:
Data collection:

Data collection was divided into four times: T0, T1, T2 and T3. T0 and T2 corresponded to preintervention data and T1 and T3 to postintervention data (T1 after the training and T3 one year later, after the whole intervention implementation).

At all four times, the I-CEpSE (competent health education practice, (in Spanish, 'Instrumento Competencia de Educación para la Salud del profesional de Enfermería'))instrument was collected as a means to measure self-reported nurses' knowledge, skills, and attitudes regarding competency-based health education. This questionnaire includes 58 items grouped into 3 domains: 1) Knowledge (items 1-23); 2) Skills (items 24-49); and 3) Attitudes (items 50-58). In turn, the skills domain is divided into two dimensions: personal/social skills (items 24-34) and educational skills (items 35-49). This is a validated instrument with good psychometric properties, internal consistency was high for each total scale (cognitive domain: Cronbach α = 0.95; psychomotor: Cronbach α = 0.95; attitudinal and affective: Cronbach α = 0.90) and for all factors (Cronbach α values ranged from 0.81-0.95).

Ethical considerations:

This study conformed to the principles set out in the Declaration of Helsinki and was approved by the centre's board and by the Research Ethics Committee (code 2019.066). Data custody complied with Organic Law 3/2018 on data protection (LOPDE). Informed consents were given to all participants. They were informed verbally and in writing about their free participation, the confidentiality and anonymity of the data and its use for scientific purposes. Nobody declined to participate or withdrew at any point of the study.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in the cardiology ward.
* Nurses working full-time and part-time.
* Nurses with permanent and temporary contracts.

Exclusion Criteria:

* Nurses who were not working during the time of the study (sick or maternity leaves).
* Nurses with short contracts (<one year).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical nurses working in the cardiology ward during the time of the intervention evaluation were the target population from which the sample was taken.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Knowledge (items 1-23), Skills: personal/social skills (items 24-34) and educational skills (items 35-49) and Attitudes (items 50-58) | T0 (2020 October)
  Measurement tool: I-CEpSE instrument
Knowledge (items 1-23), Skills: personal/social skills (items 24-34) and educational skills (items 35-49) and Attitudes (items 50-58) | T1 (2020 November)
  Measurement tool: I-CEpSE instrument
Knowledge (items 1-23), Skills: personal/social skills (items 24-34) and educational skills (items 35-49) and Attitudes (items 50-58) | T2 (2021 May first)
  Measurement tool: I-CEpSE instrument
Knowledge (items 1-23), Skills: personal/social skills (items 24-34) and educational skills (items 35-49) and Attitudes (items 50-58) | T3 (2021 May last)
  Measurement tool: I-CEpSE instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Result] Paloma B, Olano-Lizarraga M, Rumeu-Casares C, Quesada A, Saracibar-Razquin M, Vazquez-Calatayud M. [Level of empowerment of hospitalized chronic heart failure patient]. An Sist Sanit Navar. 2021 Dec 27;44(3):351-360. doi: 10.23938/ASSN.0960. Spanish. PMID 34142990
- [Derived] Vazquez-Calatayud M, Olano-Lizarraga M, Quesada-Melero AM, Rumeu-Casares C, Saracibar-Razquin M, Paloma-Mora B. Nursing capacity building in health coaching with hospitalised chronic heart failure patients: a quasi-experimental study. Contemp Nurse. 2023 Dec;59(6):443-461. doi: 10.1080/10376178.2023.2262612. Epub 2024 Jan 17. PMID 37751247
- See also: Level of empowerment of hospitalized chronic heart failure patient. — https://pubmed.ncbi.nlm.nih.gov/34142990/